CLINICAL TRIAL: NCT00672438
Title: Heritability of Opioid Effects: A Twin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Angst (Other)
Collaborators: SRI International (Industry)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SU-04212008-1119; 13018 (Other: IRB Stanford University School of Medicine)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Alfentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline placebo infusion (Placebo Comparator): Subjects will receive an intravenous infusion of normal saline.
  Interventions: Other: Saline placebo infusion
- Alfentanil infusion (Experimental): Subjects will receive an intravenous infusion of alfentanil.
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Alfentanil — Target controlled intravenous infusion of alfentanil at a plasma concentration of 100ng/ml
  Other Names: Alfenta
  Arms: Alfentanil infusion
Other: Saline placebo infusion — Intravenous infusion of normal saline
  Arms: Saline placebo infusion

SUMMARY:
Proposed twin study will test to what degree inter-individual differences in pain sensitivity and amount of pain relief in response to opioid therapy are inherited or alternatively, are due to environmental factors. This knowledge is important to guide future studies trying to explain such inter-individual differences. For example, finding that differences are largely due to environmental factors would discourage genomic studies and emphasize epidemiological studies.

DETAILED DESCRIPTION:
The principal hypothesis to be evaluated is that the degree of analgesia provided by opioids in humans displays substantial familial aggregation, and is, in fact, heritable. These studies will use a classical twin paradigm to determine the role of genetics and the environment in influencing analgesia and a range of other opioid effects.

Specific Aims: (1) Determine the degree to which opioid analgesic responses show familial aggregation and make preliminary estimates of heritability using both a heat and cold pressor pain model, and (2) determine the degree to which non-analgesic opioid responses show familial aggregation and make preliminary estimates of heritability. Side effects such as sedation, nausea, respiratory depression, and pruritus, as well as the positive affective response, a measure of abuse potential, will be monitored. Monozygotic (MZ) and dizygotic (DZ) twin pairs (125 total pairs) will be tested under controlled pain laboratory conditions for their responses to opioid infusion using the complementary pain models while monitoring side effects and additional psychometric indices of mood, sleep, and abuse potential. The selected models provide unique mechanistic information because they involve different peripheral and/or central pain pathways. DNA samples will be collected for zygosity testing and banked for future studies.

ELIGIBILITY:
Inclusion Criteria:Monozygotic or dizygotic twins ages 18-70

Exclusion Criteria:(1) Clinically relevant systemic diseases such as psychiatric, neurological, and dermatological conditions interfering with the collection and interpretation of study data (2) History of addiction (3) Allergy to study medication (4) Chronic intake of medication potentially interfering with pain processing (except oral contraceptives) (5) Intake of over-the-counter analgesics within the two days prior to study (6) Reynaud's disease (7) Pregnancy (8) Participation in other study within last 30 days (9) Personnel with direct access to addicting drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twins were recruited by a joint effort of SRI International and Stanford University School of Medicine. Initial contact and primary enrollment was the responsibility of study staff of SRI International. Recruitment was mainly achieved through the Twin Research Registry and advertisements broadcasted by regional radio stations
Pre-assignment Details: Participants were required to fast overnight except for clear liquids that were allowed up to 2 hours before starting the drug infusion. Subjects were also required to have at least 6 hours of night-time sleep before a study session.
  Some participants withdrew prior to study participation.
Groups:
- Alfentanil Infusion Prior to Saline Placebo Infusion: 50% of participants were randomized to receive an infusion of alfentanil via a computer-controlled infusion targeting steady-state plasma concentration of 100ng/ml prior to a saline placebo infusion. All other procedures were identical in both groups.
- Saline Placebo Infusion Prior to Alfentanil Infusion: 50% of participants were randomized to receive a saline placebo infusion prior to an infusion of alfentanil via a computer-controlled infusion pump targeting a steady-state plasma concentration of 100ng/ml. All other procedures were identical in both groups.
Period: Infusion 1
Arm/Group | Alfentanil Infusion Prior to Saline Placebo Infusion | Saline Placebo Infusion Prior to Alfentanil Infusion
Started | 119 | 118
Completed | 119 | 118
Not Completed | 0 | 0
Period: Washout
Arm/Group | Alfentanil Infusion Prior to Saline Placebo Infusion | Saline Placebo Infusion Prior to Alfentanil Infusion
Started | 119 | 118
Completed | 119 | 118
Not Completed | 0 | 0
Period: Infusion 2
Arm/Group | Alfentanil Infusion Prior to Saline Placebo Infusion | Saline Placebo Infusion Prior to Alfentanil Infusion
Started | 119 | 118
Completed | 119 | 118
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data collected for all enrolled participants.
Groups:
- Alfentanil Infusion Prior to Saline Placebo Infusion: 50% of participants were randomized to receive an infusion of alfentanil prior to a saline placebo infusion. All other procedures were identical in both groups.
- Saline Placebo Infusion Prior to Alfentanil Infusion: 50% of participants were randomized to receive a saline placebo infusion prior to an infusion of alfentanil. All other procedures were identical in both groups.
- Total: Total of all reporting groups
Arm/Group | Alfentanil Infusion Prior to Saline Placebo Infusion | Saline Placebo Infusion Prior to Alfentanil Infusion | Total
Number analyzed (Participants) | 122 | 120 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 120 | 242
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 46 | 46 | 92
Region of Enrollment [Number; unit: participants]
  United States | 122 | 120 | 242

OUTCOME MEASURES:

1. Primary Outcome: Heat Pain Threshold
Description: Degrees Centigrade
  Heat pain was induced with a thermal sensory analyzer (TSA-II, Medoc Advanced Medical Systems, Durham, North Carolina). A thermode was placed in contact with skin at the volar forearm. Starting at a comfortable temperature, the thermode temperature was increased at a measured rate. Study participants pushed a button of a hand-held device at the onset of pain at which point the thermode immediately reduced the temperature.
Time Frame: Participants underwent the pain testing measures at training prior to study procedures, at baseline and during each of the infusions.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: degrees centigrade
Groups:
- Alfentanil Infusion: A controlled intravenous infusion was run at a rate to target an alfentanil plasma concentration of 100ng/ml
- Saline Infusion: All participants received NS at an infusion rate identical to the alfentanil rate.
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
degrees centigrade | 49.6 [48.3 to 50.4] | 48.6 [47.1 to 49.3]

2. Primary Outcome: Cold Pain Threshold
Description: Time in seconds
  Sensitivity to cold-pressor pain was tested by asking subjects to immerse their hand up to the wrist in ice water (1-2 C) continuously re-circulated within a 12-L container with the palm of the hand in full contact with the bottom of the container.They were asked to indicate the onset of pain - reported as pain threshold.
Time Frame: as for outcome 1
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: Seconds
Groups:
- Saline Infusion: All participants received a saline infusion. All participants received NS at an infusion rate identical to the alfentanil rate.
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
Seconds | 15 [9 to 25] | 8 [6 to 13]

3. Primary Outcome: Cold Pain Tolerance
Description: Time in seconds
  Sensitivity to cold-pressor pain was tested by asking subjects to immerse their hand up to the wrist in ice water (1-2 C) continuously re-circulated within a 12-L container with the palm of the hand in full contact with the bottom of the container.They were asked to remove their hand from the water bath when it was no longer tolerable - reported as pain tolerance.
Time Frame: as for outcome 1
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
Seconds | 32 [20 to 55] | 17 [11 to 26]

4. Primary Outcome: Respiratory Rate
Description: Breaths per minute counted by direct observation and additionally recorded / external electronic monitoring.
Time Frame: Measured throughout the study session ~ 5 hours
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: Breaths per minute
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
Breaths per minute | 11 [9 to 13] | 14 [12 to 16]

5. Primary Outcome: Transcutaneous Partial Pressure of Carbon Dioxide
Description: Partial pressure of transcutaneous carbon dioxide (CO2) was measured with aid of a pO2/pCO2-electrode (Perimed Inc., North Royalton, OH) mounted to the anterior chest wall.
Time Frame: Measured continuously throughout the study session ~ 5 hours
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
mmHg | 47.7 [43.4 to 52] | 40.3 [37.6 to 42.9]

6. Secondary Outcome: Sedation
Description: Sedative opioid effects were assessed with the trail-making test (TMT) (Angst et al., 2004; Oswald and Roth, 1987). The TMT is a paper-and pencil test consisting of 4 different matrices listing numbers 1-90 in a 9 × 10 format. Subsequent numbers are located in neighboring rows or columns. Matrices were allocated randomly. Subjects had to connect numbers 1-90 as quickly as possible and the time to completion was recorded.
Time Frame: The trail making test was performed at training prior to study procedures, at baseline, and during each of the infusions.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: Time in seconds
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
Time in seconds | 70 [59 to 87] | 63 [56 to 75]

7. Secondary Outcome: Average Nausea
Description: At the end of an infusion stage participants were asked to rate the average severity of nausea on a 100-mm visual analog scale (VAS) anchored by the words "not at all" and "as much as possible." This means that the scale is 100mm long where one extreme end of the scale represents "0", and 0 represents no nausea experienced. The other extreme end of the scale represents "100", and 100 represents as much nausea as possible. Participants are asked to indicate what point on that continuum best represents their average experience.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 1 [0 to 32] | 0 [0 to 0]

8. Secondary Outcome: Maximum Nausea
Description: At the end of an infusion stage participants were asked to rate the maximum severity of nausea on a 100-mm visual analog scale (VAS) anchored by the words "not at all" and "as much as possible." This means that the scale is 100mm long where one extreme end of the scale represents "0", and 0 represents no nausea experienced. The other extreme end of the scale represents "100", and 100 represents as much nausea as possible. Participants are asked to indicate what point on that continuum best represents their maximum experience of nausea.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 8 [0 to 70] | 0 [0 to 0]

9. Secondary Outcome: Average Pruritis
Description: At the end of an infusion stage participants were asked to rate the average severity of pruritis on a 100-mm visual analog scale (VAS) anchored by the words "not at all" and "as much as possible." This means that the scale is 100mm long where one extreme end of the scale represents "0", and 0 represents no pruritis experienced. The other extreme end of the scale represents "100", and 100 represents as much pruritis as possible. Participants are asked to indicate what point on that continuum best represents their average experience of pruritis.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 20 [0 to 45] | 0 [0 to 0]

10. Secondary Outcome: Maximum Pruritis
Description: At the end of an infusion stage participants were asked to rate the maximum severity of pruritis on a 100-mm visual analog scale (VAS) anchored by the words "not at all" and "as much as possible." This means that the scale is 100mm long where one extreme end of the scale represents "0", and 0 represents no pruritis experienced. The other extreme end of the scale represents "100", and 100 represents as much pruritis as possible. Participants are asked to indicate what point on that continuum best represents their maximun experience of pruritis.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 35 [0 to 65] | 0 [0 to 0]

11. Secondary Outcome: Average Drug Liking
Description: At the end of an infusion stage participants were asked, "How much did you like the drug on average (100-mm VAS, 0 _ "not at all," 100 _ "as much as possible")? The VAS scale is 100mm long where one extreme end of the scale represents "0", and 0 indicates the participant did not like the drug experience. The other extreme end of the scale represents "100", and 100 indicates that the participant liked the drug experience as much as possible. Participants are asked to indicate what point on that continuum best represents the their experience.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 50 [0 to 75] | 0 [0 to 0]

12. Secondary Outcome: Maximum Drug Liking
Description: At the end of an infusion stage participants were asked, "What was the maximum that you liked the drug at any moment (VAS)? (100-mm VAS, 0 _ "not at all," 100 _ "as much as possible")? The VAS scale is 100mm long where one extreme end of the scale represents "0", and 0 indicates the participant did not like the drug experience. The other extreme end of the scale represents "100", and 100 indicates that the participant liked the drug experience as much as possible. Participants are asked to indicate what point on that continuum best represents the their experience.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 75 [40 to 90] | 0 [0 to 0]

13. Secondary Outcome: Maximum Drug Disliking
Description: At the end of an infusion stage participants were asked, "What was the maximum that you disliked the drug at any moment (VAS)? (100-mm VAS, 0 _ "not at all," 100 _ "as much as possible")? The VAS scale is 100mm long where one extreme end of the scale represents "0", and 0 indicates the participant did not like the drug experience. The other extreme end of the scale represents "100", and 100 indicates that the participant liked the drug experience as much as possible. Participants are asked to indicate what point on that continuum best represents the most they disliked the drug experience.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 23 [0 to 70] | 0 [0 to 0]

14. Secondary Outcome: Sedation by Patient Report
Description: Sedation was assessed by measuring cognitive speed and by asking participants to indicate on a 100-mm visual analog scale (VAS) how sedated they felt. This means that the scale is 100mm long where one extreme end of the scale represents "0", and 0 represents no sedation was experienced. The other extreme end of the scale represents "100", and 100 represents as much sedation as possible. Participants are asked to indicate what point on that continuum best represents their experience of sedation.
Time Frame: At the end of each infusion stage. 2 times total.
Population: All participants were included for analysis.
Measure: Median (Inter-Quartile Range); unit: numerical score
Arm/Group | Alfentanil Infusion | Saline Infusion
Number analyzed (Participants) | 228 | 228
numerical score | 75 [60 to 87] | 0 [0 to 15]

ADVERSE EVENTS:
Time Frame: Baseline to conclusion of study session (+/- 5 hours).
Description: Participant vital signs, including respiratory rate, CO2 levels, oxygen saturation, ECG, pulse rate, and level of consciousness were measured throughout the study session.
Groups:
- Alfentanil: Intravenous infusion of Alfentanil
Arm/Group | Alfentanil
Serious Adverse Events (participants affected / at risk) | 0/228
Other Adverse Events (participants affected / at risk) | 0/228

LIMITATIONS AND CAVEATS:
The study was completed as intended, enrolling 121 twin pairs for a total of 114 evaluable pairs. There are no unexpected adverse events to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No